CLINICAL TRIAL: NCT05732168
Title: A Test Battery for Evaluation of Muscle Strength, Balance and Functional Performance in Subjects With Chronic Ankle Instability: a Cross-sectional Study
Brief Title: A Test Battery for Evaluation of Muscle Strength, Balance and Functional Performance in Subjects With Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Ryman Augustsson, Associate Professor, Linnaeus University
Other Study IDs: EPK 676 - 2021
Record Dates: First submitted 2023-01-24; First posted 2023-02-16 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with chronic ankle instability: Men and women with recurrent unilateral ankle instability problems
  Interventions: Diagnostic Test: A test battery for evaluation of muscle strength, balance and functional performance
- Control group: Healthy men and women without ankle problems
  Interventions: Diagnostic Test: A test battery for evaluation of muscle strength, balance and functional performance

INTERVENTIONS:
Diagnostic Test: A test battery for evaluation of muscle strength, balance and functional performance — Subjects with chronic ankle instability (CAI) were evaluated with five tests of strength, balance and functional performance.

SUMMARY:
Purpose: The primary aim of this study was to investigate subjects with chronic ankle instability regarding strength, balance and functional performance with an easily used test battery that required minimal equipment. A second aim was to evaluate which of these tests that has the highest ability to discriminate impaired function between injured and non-injured ankle in CAI subjects.

Methods: This study was conducted with a cross-sectional design. A total of 20 (11 women) CAI subjects, engaged in sports, were tested for assessment of strength, balance and functional performance using the following tests; isometric strength in inversion and eversion, the single leg stance test (SLS), single leg hop for distance (SLHD) and side hop test. Additionally, 15 healthy subjects were tested with the same test battery for the evaluation of

DETAILED DESCRIPTION:
Study design and procedure Data for cross-sectional study, adhering to the STROBE statement were collected during 2021-2022 where subjects with chronic ankle instability (CAI) were evaluated with tests of strength, balance and functional performance.

Outcome measures The primary outcome was ankle function, in subjects with CAIs, which was assessed by a test battery consisting of two muscle strength tests, one balance test and two functional performance tests.

Muscle strength Ankle inversion and eversion isometric muscle strength were assessed using hand-held dynamometry, MicroFET2 (Hoggan Health Industries, Inc., Draper, UT). The subjects were examined in a lying in a prone position with the feet outside the edge with one test leader stabilizing the subject's lower leg. Before the test, the subjects tried the directions against the test leader's hand. Three maximal isometric contractions, measured in Newton (N) with 15 secs of rest between each contraction, were measured and the best attempt was used for further analysis. Five minutes of rest was used when changing test direction.

The single leg stance test (SLS) Balance was measured with the Single-leg stance test (SLS). The test began with the subject standing on one leg, with his arms straight down, and the other leg held against the calf of the standing leg. When standing steadily, the subject was asked to close their eyes and maintain balance without using opposite legs or arms. The number of times the subject corrected his balance, during 30 sec, was documented as part foot lifts. Part foot lift was defined as all parts of the foot that left the surface, e.g. toes, outside foot, heel. Putting down the opposite leg also counted as part foot lift. The total number of part foot lifts constituted a score that was used as a result.

Functional performance Functional performance was assessed by the Single-leg hop for distance (SLHD) and the 30-sec timed side hop test. Before each test, the subject had to perform three submaximal test jumps.

For the SLHD, the subject was standing on one leg with the other leg lifted from the floor. Free leg swing was allowed but the hands was placed behind the back. The subject jumped forward as far as possible, taking off and landing on same foot with a controlled landing. The subject had to maintain balance on landing until the test leader had registered the landing position, approximately (2-3 s). The distance was measured in centimeters from the toe at the push-off to the heel where the subject landed.

For the side hop test, the subject stood on the test leg, with the other leg lifted from the floor, and hands placed behind the back. Two parallel strips of tape, placed 40 cm apart on the floor was used and the subject jumped from side to side as many times as possible during a period of 30 s. The number of successful jumps performed, without touching the tape, was recorded and will be used for further analysis.

Sample size calculation Based on a power of 0.80 (α =0.05), approximately 18 CAI subjects would be required to detect a 20 % difference between injured and non-injured ankle in the balance test score. Twenty percent was considered as a minimal clinically relevant difference. Therefore, this study was planned to recruit a minimum of 25 CAI subjects with regard for potential dropouts.

Statistical analysis plan Statistics will be calculated using IBM SPSS (IBM SPSS Statistics for Windows, Version 27.0. IBM, Armonk, NY). Differences in strength, balance and functional performance, between injured and non-injured ankle, will be analyzed with the Wilcoxon rank test. The Spearman's correlation coefficient will be used to analyze the association between the different tests.

The limb symmetry index (LSI) will be calculated to determine whether a side-to-side lower limb difference could be classified as normal or abnormal. The LSI is defined as the ratio of the score of the injured ankle and the score of the non-injured ankle, expressed in percent (injured/non-injured x 100 = LSI).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ankle problems
* Aged 15-40 years
* Minimum three recurrent sprains in the past year

Exclusion Criteria:

* previous ankle fracture with internal fixation surgery
* disease / illness that could have a general effect on the balance or strength
* newly sprained/injured in the current ankle within a period of eight weeks before the test

Ages: 15 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 27 CAI received an invitation to participate. Four subjects were excluded due to newly injured ankle, two due to bilateral ankle instability and one because of previous problems but not in the past year. Finally, 20 CAI subjects were included in the analysis (Table 1). The subjects were involved in floorball (n=8), running (n=5), football (n=5), equestrian sports (n=1) and gymnastics (n=1). In addition, a convenience sample of 15 healthy subjects were also recruited in order to establish the specificity and accuracy of the test battery.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Muscle strength measured in Newton | 1 day
  Ankle inversion and eversion isometric muscle strength measured with a handheld dynometer and measured in Newton
Balance | 1 day
  Balance assessed by the Single-leg stance test (SLS) and measured in number of footlifts
Functional performance assessed with the SLHD test measured in centimeters | 1 day
  Functional performance assessed with the SLHD test measured in centimeters for the total distance. The athlete stands on one leg and then jump as far as possible and land on the same leg. The best of three attempts will be used for further analysis.
Functional performance assessed with the side hop test and measured as the number of repetitions | 1 day
  Functional performance assessed with the side hop test and measured as the number of repetitions. Two parallel strips of tape is placed 40 cm apart on the floor. The athlete stands on one leg, with the hands behind the back, and jumps from side to side between the two strips. The athlete jumps as many times as possible during a period of 30 s. The number of successful jumps performed, without touching the tape, is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryman Augustsson S, Sjostedt E. A test battery for evaluation of muscle strength, balance and functional performance in subjects with chronic ankle instability: a cross-sectional study. BMC Sports Sci Med Rehabil. 2023 Apr 13;15(1):55. doi: 10.1186/s13102-023-00669-5. PMID 37055818